CLINICAL TRIAL: NCT06181526
Title: The Study of Safety and Preliminary Efficacy of Aleeto in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Safety and Preliminary Efficacy of Aleeto in Amyotrophic Lateral Sclerosis
Acronym: SPECIALS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Vice President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: KY2023-252-01
Record Dates: First submitted 2023-12-06; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Placebo parallel-controlled; Single-center Study; Double Blind Study; Randomized Controlled Trial; Dose escalation clinical study; Aleeto
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Injections, Intravenous; Injections, Spinal

STUDY DESIGN:
Intervention Model Description: In this study, a dose-escalation clinical trial is conducted to explore the maximum tolerated dose, and three dose groups are set: 0.5 μg/kg, 1 μg/kg, and 2 μg/kg, with 3 cases in the initial dose group and placebo group, and 6 cases in the follow-up dose group, with a total of 24 subjects.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intrathecal administration combined with intravenous administration of Aleeto(0.5μg/kg) or placebo (Experimental): Four patients will be randomly assigned to the treatment group and the placebo group. 3 patients will receive intrathecal administration combined with intravenous administration of 0.5 μg/kg Aleeto and sodium chloride, while another patient will receive the same dose of placebo.
  Day 1-12: Intrathecal administration of Aleeto will be conducted on Days 1, 4, 8, and 11, and intravenous administration of Aleeto on Days 2, 3, 5, 6, 9, 10, 12, and 13.
  Day 31-36: Intrathecal administration of Aleeto will be conducted on Days 31 and 34, and intravenous administration of Aleeto on Days 32, 33, 35, and 36.
  D61-66: Intrathecal administration of Aleeto will be conducted on Days 61 and 64, and intravenous administration of Aleeto on Days 62, 63, 65, and 66.
  Interventions: Drug: Aleeto; Device: intravenous injection; Device: intrathecal injection
- Intrathecal administration combined with intravenous administration of Aleeto (1μg/kg) or placebo (Experimental): Seven patients will be randomly assigned to the treatment group and the placebo group. 6 patients will receive intrathecal administration combined with intravenous administration of 1μg/kg Aleeto and sodium chloride, while another patient will receive the same dose of placebo.
  Day1-12: Intrathecal injection of Aleeto would be given on Day 1, 4, 8, and 11, and intravenous injection of Aleeto on Day 2, 3, 5, 6, 9, 10, 12, and 13.
  Day31-36: Intrathecal injection of Aleeto would be given on Day 31 and 34, and intravenous injection of Aleeto on Day 32, 33, 35, and 36.
  D61-66: Intrathecal injection of Aleeto would be given on Day 61 and 64, and intravenous injection of Aleeto on Day 62, 63, 65, and 66.
  Interventions: Drug: Aleeto; Device: intravenous injection; Device: intrathecal injection
- intrathecal injection and intravenous injection of Aleeto (2μg/kg) or placebo (Experimental): Seven patients will be randomly assigned to the treatment group and the placebo group. 6 patients will receive intrathecal administration combined with intravenous administration of 2μg/kg Aleeto and sodium chloride, while another patient will receive the same dose of placebo.
  Day1-12: Intrathecal injection of Aleeto would be given on Day 1, 4, 8, and 11, and intravenous injection of Aleeto on Day 2, 3, 5, 6, 9, 10, 12, and 13.
  Day31-36: Intrathecal injection of Aleeto would be given on Day 31 and 34, and intravenous injection of Aleeto on Day 32, 33, 35, and 36.
  D61-66: Intrathecal injection of Aleeto would be given on Day 61 and 64, and intravenous injection of Aleeto on Day 62, 63, 65, and 66.
  Interventions: Drug: Aleeto; Device: intravenous injection; Device: intrathecal injection
- intravenous injection of Aleeto (2μg/kg) (Experimental): Six patients will receive intravenous administration of 2 μg/kg Aleeto and sodium chloride.
  Day1-12: Patients would be given intravenous injection of Aleeto(2μg/kg) +100ml sodium chloride for 12 days (Day 1 to 6, 8 to 13) once a day.
  Day31-36: Patients would be given intravenous injection of Aleeto(2μg/kg) +100ml sodium chloride for 6 days (Day 31 to 36) once a day.
  D61-66: Patients would be given intravenous injection of Aleeto(2μg/kg) +100ml sodium chloride for 6 days (Day 61 to 66) once a day.
  Interventions: Drug: Aleeto; Device: intravenous injection

INTERVENTIONS:
Drug: Aleeto — According to the groups, patients would be treated with Aleeto via intrathecal injection or intravenous injection, and the specific dosage and administration method of Aleeto will depend on the grouping.
Device: intravenous injection — According to the groups, patients would be treated with Aleeto or placebo +100ml sodium chloride injection via intravenous injection, depend on the grouping
Device: intrathecal injection — According to the groups, patients would be treated with Aleeto or placebo + 8ml sodium chloride injection via intrathecal injection, depend on the grouping.
  Arms: Intrathecal administration combined with intravenous administration of Aleeto (1μg/kg) or placebo; Intrathecal administration combined with intravenous administration of Aleeto(0.5μg/kg) or placebo; intrathecal injection and intravenous injection of Aleeto (2μg/kg) or placebo

SUMMARY:
This study is a single-center, randomized, double-blind, placebo parallel-controlled, dose-escalation clinical study. The aim of this study was to evaluate the safety, tolerability, and preliminary effect of Aleeto in adult patients with ALS, and to provide an appropriate dose for the future clinical trial.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a fatal neurodegenerative disease, which is characterized by progressive loss of number and function of upper and lower motor neurons located in the brain and spinal cord, which leads to paralysis. ALS mainly begins in the limbs and face, where about one-third of patients have difficulty in speaking, chewing, or swallowing, then progressively affecting the pharyngeal muscles, attacking the sphincter in the advanced stages of the disease, and eventually affecting the trunk and respiratory function as the disease progresses.

"Aleeto" derived from cellular exosomes, is a group of specific microenvironment protein polymers secreted by stem cells under stressed conditions, which has the advantages of selective assembly, targeted delivery, efficient repair of damaged tissues, high safety, stable chemical properties, and easy preservation. What's more, Aleeto has a strong nerve repair function.

This study is a single-center, randomized, double-blind, placebo parallel-controlled, dose-escalation clinical study, aiming to evaluate the safety, tolerability, and preliminary effect of Aleeto in adult ALS patients, and provide an appropriate dose for the future clinical trial.

In this study, we plan to enroll 24 patients, and will be randomly assigned to 4 groups. The initial dose group consists of four subjects, out of which three subjects will receive intravenous administration and intrathecal administration of 0.5μg/kg Aleeto, while one subject will receive a placebo. Fourteen subjects will be randomly assigned to the 1μg/kg and 2μg/kg dose groups to receive intrathecal administration combined with intravenous administration, with one subject in each dose group randomly receiving placebo treatment. Six subjects will be randomly assigned to the 2μg/kg dose group to receive intravenous administration only. Data are collected in face-to-face interviews at baseline and Day 14, 30, 37, 60, 67, 90, 120 follow-up visits. All patients will be examined before and after treatment, and the results will be compared.

The primary outcomes are the incidence of adverse events (AEs) and serious adverse events (SAEs), and the incidence of abnormal changes in laboratory examination indicators, vital signs, neurological physical examination, and electrocardiogram within 120 days after the treatment. The secondary outcomes included changes in immunological indicators, pharmacokinetics, ALS Functional Rating Scale-Revised (ALSFRS-R), as well as the incidence of invasive mechanical ventilation and mortality rate .

The statistical analysis was performed by bilateral test, and the test level α was 0.05.

Baseline Equilibrium Analysis: Analysis of variance or Kruskal-Wallis H test is used to compare continuous data.The Chi-Squared test or Fisher's exact test is used to compare the categorical data.

Primary Efficacy Analysis: The comparability among different dosage groups in terms of incidence of adverse events (abnormal liver functions, hypersensitivity reactions, liver failure, dyspnea, etc.), severe adverse events, and other abnormal indicators will be analyzed using Chi-squared tests or Fisher's exact test. Changes in laboratory examination indicators and vital signs before and after treatment will be analyzed using paired t-tests or Wilcoxon signed rank sum test. The intergroup differences in laboratory examination indicators and changes in vital signs before and after treatment will be analyzed using t-test or Mann-Whitney U test.

Secondary Efficacy Analyses: The improvement of immunological indicators (lymphocyte subgroup analysis), pharmacokinetic indicators, and ALSFRS-R before and after treatment will be analyzed using paired t-tests or Wilcoxon signed rank sum test. The intergroup comparison of immunological indicators (lymphocyte subgroup analysis), pharmacokinetic indicators, and ALSFRS-R before and after treatment will be analyzed using t-tests or Mann-Whitney U tests. The intergroup significance of the incidence of invasive mechanical ventilation and mortality rate is determined using Chi-squared tests or Fisher's exact test.

Exploratory Analysis: Comparison of measurement data: The improvement of ALSAQ-40, EQ-5D-5L, modified Norris scale, forced lung capacity, muscle strength, electromyographic indicators, gait function, biomarker levels, FSS, imaging indicators, HAMA and HAMD scales will be analyzed using paired t-tests or Wilcoxon signed rank sum test. The above exploratory analysis indicators and the difference in survival time between two groups will be analyzed using t-test or Mann-Whitney U test. Analysis of variance or Kruskal Wallis H-test will be used for comparing the differences ａｍｏｎｇ different dosａｇｅ groups, and Bonferroni correction method will be used for multiple comparisons. Mixed linear models will be used for analyzing the differences in the trend of changes between different dose groups over a period of 120 days (the data which corresponds to skewed distribution will be transformed). LSmeans will be used for analyzing the differences of indicators between different groups at different times, as well as the differences within the same group at different times.

Comparison of enumeration data: Chi-square test or Fisher's exact test for enumeration data.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are qualified for the clinical trial program cycle judged by well-trained physicians;
2. 18 years old≤ age≤ 75 years old, males or females;
3. Forced vital capacity ≥ 80% of predicted vital capacity during the screening period;
4. The total score of the ALSFRS-R scale ≥ 30 points and ≤40 points during enrollment, and the respiratory function item ≥ 3 points;
5. Diagnosis of confirmed or probable ALS in accordance with the revised EI Escorial diagnostic criteria for amyotrophic lateral sclerosis of the World Federation of Neurology;
6. Subjects or their legal representatives clearly understand and voluntarily participate in the study and sign the informed consent form;
7. Subjects (including male subjects) are willing to have no birth plan and voluntarily take effective contraceptive measures during the entire study period and within 3 months after the end of the study, and have no plan to donate sperm or eggs.

Exclusion Criteria:

1. Diagnosed with familial ALS (based on family history);
2. With obvious cognitive impairment (MMSE scale: ≤19 points in the illiteracy group，≤ 22 points in the primary school group, and ≤26 points in the junior high school group (more than 8 years of education);
3. Obvious dysphagia;
4. Positive HIV test or history of positive test;
5. Positive hepatitis C virus antibody or positive test history;
6. Hepatitis B active infection (hepatitis B surface antigen positive and/or serum HBV DNA positive or serum HBV DNA > 2 × 108 IU/ml;
7. Have used other investigational drugs within 1 month or within 5 drug half-lives;
8. Diseases and deformities of the lumbar spine;
9. Have other conditions known to be associated with motor neuron dysfunction that may confuse or obscure an ALS diagnosis;
10. Other psychiatric disorders diagnosed according to DSM-V diagnostic criteria, or significant suicide intent;
11. With severe hepatic insufficiency, renal insufficiency or severe cardiac insufficiency (severe hepatic insufficiency refers to ALT value≥2.0 times the upper limit of normal value or AST value≥2.0 times the upper limit of normal value; severe renal insufficiency refers to CRE≥1.5 times the upper limit of normal value or eGFR<40mL/min/1.73m2; severe cardiac insufficiency refers to NYHA class 3-4);
12. Permanently dependent on ventilator-assisted ventilation;
13. History of alcohol and drug abuse; Edaravone users;
14. Patients who are pregnant, breast-feeding, or who are likely to become pregnant and plan to become pregnant;
15. Patients participating in other clinical trials or using other biological agents, drugs, or devices under investigation;
16. Patients who have received any vaccinations within 28 days;
17. Contraindications to MRI (eg, claustrophobia);
18. Unable to be cooperative and complete the follow-up due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events and serious adverse events (SAEs) | from Day 1 to Day 120
  Close monitoring of patients for any physical discomfort, such as shortness of breath, rash, etc. Regular follow-up examinations of liver function, kidney function, blood routine, and other laboratory parameters should be performed. Adverse events includes abnormal liver biochemical indicators, hypersensitivity, liver failure, dyspnea, etc.
Incidence of changes in clinical laboratory examination indicators, changes in vital signs, abnormal neurological examination and abnormal electrocardiogram | from Day 1 to Day 120
  After Aleeto treatment in adult patients with ALS, monitor patients' blood routine, biochemistry, vital signs, electrocardiogram, physical examination, and other parameters.

SECONDARY OUTCOMES:
Immunological markers | Day 2, Day 7, Day 14, Day 30, Day 32, Day 37, Day 60, Day 62, Day 67, Day 90, Day 120
  After Aleeto treatment in adult patients with ALS, regular reevaluation of patients' lymphocyte subpopulations.
Time to invasive mechanical ventilation and death | Day 2, Day 7, Day 14, Day 30, Day 32, Day 37, Day 60, Day 62, Day 67, Day 90, Day 120
  After Aleeto treatment in adult patients with ALS, record the time of respiratory distress requiring the use of a ventilator and the time of death.
Pharmacokinetics analysis | Day 1, Day 6, Day 13, Day 31, Day 36, Day 61, Day 66
  Blood samples will be collected at 1 hour, 2 hours, 4 hours, and 6 hours after administration to test the half-life period of Aleeto.
Pharmacokinetics analysis | Day 1, Day 6, Day 13, Day 31, Day 36, Day 61, Day 66
  Blood samples will be collected at 1 hour, 2 hours, 4 hours, and 6 hours after administration to test the peak time of Aleeto.
Pharmacokinetics analysis | Day 1, Day 6, Day 13, Day 31, Day 36, Day 61, Day 66
  Blood samples will be collected at 1 hour, 2 hours, 4 hours, and 6 hours after administration to test the maximum plasma concentration of Aleeto.
ALS Functional Rating Scale-Revised | Day 120
  Complete the ALS Functional Rating Scale-Revised scale assessment again 120 days after enrollment, which score is range from 0 to 48, and lower scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, MD+PhD, Principal Investigator — Capital Medical University
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No